CLINICAL TRIAL: NCT06879808
Title: The Effect of Color Therapy on Depression, Stress, Anxiety and Quality of Life in Hemodialysis Patients: A Randomized Controlled Study
Acronym: Color Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Safiye Yanmış, Assistant Professor, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Erzi̇ncanBinaliYildirimUni; Scientific Research Projects (Other Grant/Funding Number: Fırat University)
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hemodialysis; Color Therapy
Keywords: Anxiety; Color Therapy; Depression; Hemodialysis; Nursing; Quality of Life; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Color Therapy

STUDY DESIGN:
Intervention Model Description: Randomization; participants were divided into two groups by using simple random numbers table, and then the first group which was drawn by lot method was named as the experimental group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Color therapy group (Experimental): group doing color therapy
  Interventions: Other: Color therapy
- No color therapy group (No Intervention): group not doing color therapy

INTERVENTIONS:
Other: Color therapy — In the experimental group, color therapy was applied 3 days a week for the first two weeks, while no intervention was performed in the third and fourth weeks. In the fifth and seventh weeks, color therapy was applied for 15 minutes each day, while no intervention was performed in the sixth week.
  Arms: Color therapy group

SUMMARY:
This study was conducted to examine the effect of color therapy on depression, stress, anxiety and quality of life in hemodialysis patients.

DETAILED DESCRIPTION:
Many patients on hemodialysis treatment require hemodialysis, which requires hospitalization three times a week for four hours each dialysis session. Therefore, practices such as color therapy may be useful in the management of psychological symptoms in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Be on hemodialysis treatment for at least 6 months,
* No sleeping pills or sedative medication,
* No physical or cognitive impairment that prevents them from understanding the education and no diagnosis of a psychiatric illness,
* The patient or someone living in the same household with the patient is literate,
* Patients have no vision problems,
* Patients must be 18 years of age or older.

Exclusion Criteria:

* Being on hemodialysis treatment for less than 6 months,
* Taking sleeping pills or sedative medication,
* Being diagnosed with a physical illness or cognitive impairment or psychiatric illness that prevents understanding the education provided,
* Illiteracy of the patient and relatives,
* Patients have vision problems,
* Refusing to participate in the research,
* Under 18 years of age

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress-21 scale (DASS-21) | 8 week
  The 21-question DASS scale used in the study was taken by Henry and Crawford. This scale (DASS-21) has 7 questions each to measure the dimensions of depression, stress and anxiety. The scale is a 4-point Likert-type scale, coded as 0 "not applicable to me", 1 "somewhat applicable to me", 2 "generally applicable to me", and 3 "completely applicable to me".
Short Form-12 (SF-12) Quality of Life Scale | 8 week
  Ware et al. decided to develop a more practical form of the SF-36 that could be administered in a shorter time and developed the SF-12, which contains the same sub-dimensions as the SF-36 by reducing the number of questions. In addition to the fact that the SF-12 was created in such a way that the same component summary scores can be obtained as the SF-36, the fact that it contains fewer items and therefore has a shorter administration time provides a great advantage. Although it has been demonstrated that the SF-36 scale has sufficient validity and reliability in studies conducted in both patient and normal sample groups in our country, the validity and reliability study of the Turkish form of the SF-12, which was developed as a shorter alternative to the SF-36, was attempted. Similar to SF-36, SF-12 consists of 8 sub-dimensions and 12 items including physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social function

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bahçecioğlu Turan, Associate Professor, Principal Investigator — Firat University; Zülfünaz Özer, Associate Professor, Study Director — Istanbul Sebahattin Zaim University; Safiye Yanmış, Assistant Professor, Study Director — Erzincan Binali Yildirim Universitesi; Mukadder Mollaoğlu, Professor Doctor, Study Director — Cumhuriyet University
Locations (1):
- Fırat University, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the article is published